CLINICAL TRIAL: NCT04404647
Title: Irreversible Electroporation of Unresectable Liver Tumors - a Phase I Study of Safety and Feasibility
Brief Title: Irreversible Electroporation of Unresectable Liver Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor of surgery, Consultant surgeon, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20190072
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Liver Metastases; Hepatocellular Carcinoma; Bile Duct Cancer
Keywords: irreversible electroporation; primary liver cancer; secondary liver cancer; colorectal liver metastases; NanoKnife; ablation; IRE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Selected patients who choose to participate will undergo ablation of the target lesion using irreversible electroporation.
  Interventions: Procedure: Irreversible electroporation

INTERVENTIONS:
Procedure: Irreversible electroporation — The IRE procedure will be carried out as ultrasound guided technique either percutaneously or during laparotomy. Needle spacing and electrical pulse delivery will be performed in a standardized way.
  Other Names: NanoKnife(TM)

SUMMARY:
The aim of this study is to evaluate the safety and feasibility of curative intended irreversible electroporation (IRE) in the treatment of liver tumors neighboring major vessels or bile ducts.

DETAILED DESCRIPTION:
Patients can be included in the study if they have one or more malignant liver tumors unsuitable for resection and thermal ablation (due to proximity of major vessels or bile duct) or other established liver directed therapies.

Prior to inclusion all potential participant will be evaluated by the local multidisciplinary team, to insure fulfillment of the above-mentioned criteria. In general, the included patient will have tumors with <1 cm of margin to major hepatic vessels or bile ducts, thereby not allowing for conventional treatments because of risk of i.e. hemorrhage, biliary tract damage, liver failure or ineffective ablation due to heat sink.

IRE will be done under general anesthesia as an in-patient procedure. Patients will be observed for at least 24 hours after IRE.

Patients will attend CT scans 1, 3, 6, 9, 12, 18, 24, 36, 48 and 60 months post-IRE according to national guidelines (for follow-up after radiofrequency ablation (RFA)). Patients will attend the out-patient clinic after 1, 3, 6, 9, 12, 18 and 24 months. During the follow-up period, patients will be asked to fill out electronic forms monitoring pain, quality of life and nutritional status. After 24 months the patients will only be followed with CT scans in accordance with the mentioned schedule. Data collection for scientific purposes will stop when the last included patient has been followed for at least 24 months or when the study period concludes.

In case of multiple liver tumors, where a conventional treatment approach is not possible due to a single lesion being too close to major vessels or bile ducts, IRE may be used in conjunction to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary cancer of the liver.
* Largest tumor diameter ≤5 cm in any plane.
* Tumor must be deemed as unresectable and unsuitable for other established curative liver directed therapies.
* Treatment must be given with curative intent.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Radiological signs of synchronous intra- or extrahepatic disease, unless curative intended therapy is planned.
* Tumor is inaccessible e.g. due to venous dilation etc. (assessed with preoperative ultrasound)
* American Society of Anesthesiologists (ASA) score >3
* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Child-Pugh class C
* International Normalized Ratio (INR)>1.5
* Pregnancy
* Persistent atrial fibrillation
* Implanted electronic devices e.g. cardiac pacemakers or other electrostimulators.
* Metal stents or other metallic objects near the ablation zone (unless the stent can be replaced with a plastic stent prior to IRE)
* Severe allergies to anesthetic agent, paralytic agent or any of the equipment used during treatment.
* Patient is referred from a hospital outside of Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
90-day complication rate and severity | 90 days after intervention (last patient)
  Adverse events will be registered and scaled according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Technical success rate | 90 days after intervention (last patient)
  The rate of patients were it is possible to place needles according to the treatment plan and deliver 90 electrical pulses per electrode pair
Technical efficacy rate (1 month) (according to SIR) | 90 days after intervention (last patient)
  The rate of patients showing no residual tumor on contrast enhanced computed tomography (ceCT)
Median local progression free survival from IRE | 2 years after intervention (last patient)
  The median time from the intervention to progressive disease of the treated lesion, according to RECIST 1.1 or modified RECIST (mRECIST) (only for HCC).
Median overall survival (OS) from IRE | 2 years after intervention (last patient)
  The median time from the intervention to death.
Longitudinal changes in perceived quality of life | 2 years after intervention (last patient)
  Quality of life questionnaire - Core 30 is used to assess the quality of life in the included patients. Raw scores will be calculated according to the manual. Items will be grouped in: Global health status (range 0 - 100, high is good), Functional scales (range 0 - 100, high is good) and symptom scales (range 0 - 100 low is good). Differences in each scales during the course of the trial will be calculated separately.
Longitudinal changes in pain perception | 2 years after intervention (last patient)
  Long term pain will be assessed using the modified Danish version of the Brief Pain Inventory - short form. The outcomes assessed will be an average score of pain severity items and interference items in accordance with the manual. The scales range from 0 to 10 (lower is less pain).
Periprocedural pain perception | 90 days after intervention (last patient)
  Perioperative pain will be scores using the visual analogue pain scale (range 0 - 10, low score is less pain).
Longitudinal changes in Eastern Cooperative Oncology Group (ECOG) performance status | 2 years after intervention (last patient)
  Physicians assessment of global functioning using the "Eastern Cooperative Oncology Group" performance status scale (range 0 - 5, low score is better)
Longitudinal changes in nutritional status assessment | 2 years after intervention (last patient)
  Nutritional status assessment using the Scored Patient-Generated Subjective Global Assessment (short form). The short form includes only patient reported measures and will be combined into a single score according to the manual (range 0 - 37, low score is better).

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, DMSc, Study Director — Department of Gastrointestinal Surgery, Aalborg University Hospital
Locations (1):
- Department of Gastrointestinal Surgery, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No